CLINICAL TRIAL: NCT01028053
Title: A Principal Open-label Study to Assess the Prognostic Usefulness of Flutemetamol (18F) Injection for Identifying Subjects With Amnestic Mild Cognitive Impairment Who Will Convert to Clinically Probable Alzheimer's Disease
Brief Title: Assess the Prognostic Usefulness of Flutemetamol (18F) Injection for Identifying Subjects With Amnestic Mild Cognitive Impairment Who Will Convert to Clinically Probable Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: Medpace, Inc. (Industry); i3 Statprobe (Industry); i3 Research (Industry); Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-067-005
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
Keywords: Mild Cognitive Impairment; Positron Emission Tomography; National Institute of Neurological and Communicative Disorders and Stroke; Alzheimer's Disease and Related Disorders Association; Assess Prognostic Usefulness of Flutemetamol Injection for Identifying Subjects who will Convert to Clinically Probable Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Communication Disorders; Stroke | interventions — flutemetamol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Flutemetamol (18F) Injection (Experimental): Flutemetamol (18F) Injection
  Interventions: Drug: Flutemetamol (18F) Injection

INTERVENTIONS:
Drug: Flutemetamol (18F) Injection — All subjects will receive an i.v. dose of (18F) flutemetamol (less than 10 mg flutemetamol). The nominal activity of a single administration of (18F) flutemetamol will be 185 MBq.
  Other Names: Flutemetamol; 18F

SUMMARY:
This study will investigate the efficacy of the Flutemetamol (18F) Injection PET tracer in identifying abnormal (18F) flutemetamol uptake patterns which predict the conversion from aMCI to a b-amyloid associated clinically probable Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 60 years old or older.
* The subject meets the Petersen criteria for amnestic MCI.
* The subject has a score of less than or equal to 4 on the Modified Hachinski Ischemic Scale.
* The subject has a MMSE score of 24-30.
* The subject has a non-contrast MRI examination as part of the screening visit that excludes aMCI arising from structural causes.
* The subject and/or the subject's legally acceptable representative, if applicable, in accordance with local regulations, has signed and dated an informed consent.

Exclusion Criteria:

* The subject has any significant neurologic disease other than suspected aMCI; such as Parkinson's disease, Huntington's disease, normal pressure hydrocephalus, brain tumor, supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits, or known structural brain abnormalities.
* The subject has one or more aneurysm clips, artificial heart valves, metal implants, embedded metal fragments or pacemakers that would pose a risk during an MRI.
* The subject has major depression, bipolar disorder, as described in the DSM-IV within the past year.
* The subject has history of schizophrenia (DSM-IV criteria).
* The subject has had, within the prior 3 months, psychotic features, agitation or behavioral problems that could lead to protocol compliance issues.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2009-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sherwin, M.D., Study Chair — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

REFERENCES:
- [Derived] Pichet Binette A, Palmqvist S, Bali D, Farrar G, Buckley CJ, Wolk DA, Zetterberg H, Blennow K, Janelidze S, Hansson O. Combining plasma phospho-tau and accessible measures to evaluate progression to Alzheimer's dementia in mild cognitive impairment patients. Alzheimers Res Ther. 2022 Mar 29;14(1):46. doi: 10.1186/s13195-022-00990-0. PMID 35351181

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flutemetamol (18F) Injection
Started | 365
Completed | 232
Not Completed | 133
Not completed — Screen Failure | 113
Not completed — Patient Request | 11
Not completed — Protocol Violation | 1
Not completed — Physician Decision | 2
Not completed — Technical Problem | 1
Not completed — Terminated by Sponsor | 1
Not completed — Various reasons | 4

BASELINE CHARACTERISTICS:
Arm/Group | Flutemetamol (18F) Injection
Number analyzed (Participants) | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (8.62)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 63
  >=65 years | 169
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118
  Male | 114
Region of Enrollment [Number; unit: participants]
  United States | 109
  Belgium | 13
  Denmark | 8
  Finland | 15
  Sweden | 7
  United Kingdom | 80

OUTCOME MEASURES:

1. Primary Outcome: Hazard Ratio (HR) by PET Scan Readers for Conversion to Probable Alzheimer's Disease Based on Visual Image Interpretation.
Description: Visual Interpretation of the PET scan by independent readers.
  Note: The statistic Hazard ratio (HR) is the ratio of the hazard rates in the 2 groups (1 group being normal (negative for amyloid B) and 1 group being abnormal (positive for amyloid B). Under the null hypothesis of equal rates, the HR would be equal to 1.
  As the HR increases above 1, the chances of being probable Alzheimer's Disease (pAD) also increases.
  Note: Eight Subjects who withdrew prior to the first Clinical Adjudication Committee (CAC) evaluation are not included in the analysis. (232 - 8 = 224 Subjects included).
Time Frame: Up to 36 months post flutemetamol administration
Population: Eight Subjects who withdrew prior to the first Clinical Adjudication Committee (CAC) evaluation are not included in the analysis. (232 - 8 = 224 Subjects included).
Measure: Number; unit: Ratio of visual interpretations
Groups:
- Hazard Ratio: The statistic Hazard ratio (HR) is the ratio of the hazard rates in the 2 groups (1 group being normal (negative for amyloid B) and 1 group being abnormal (positive for amyloid B). Under the null hypothesis of equal rates, the HR would be equal to 1.
  As the HR increases above 1, the chances of being probable Alzheimer's Disease (pAD) also increases.
Arm/Group | Hazard Ratio
Number analyzed (Participants) | 224
Ratio of visual interpretations
  Reader 1 - Visual Interpretation | 3.418
  Reader 2 - Visual Interpretation | 1.962
  Reader 3 - Visual Interpretation | 2.561
  Reader 4 - Visual Interpretation | 2.633
  Reader 5 - Visual Interpretation | 2.580

2. Secondary Outcome: The of Normal and Abnormal Subjects Who Convert to Probable Alzheimer's Disease (pAD) Within the Follow up Period.
Description: Numbers of subjects with normal and abnormal patterns of [18F]flutemetamol uptake who converted to pAD.
Time Frame: Up to 36 months post flutemetamol administration.
Population: as for outcome 1
Measure: Number; unit: Number of subjects
Groups:
- Not Clinically Probable Alzheimer's Disease: A blinded visual interpretation of a clinical diagnosis of the number of Normal-Scan and Abnormal-Scan Subjects who Converted to not clinically probable Alzheimer's Disease (pAD).
- Clinically Probable Alzheimer's Disease: A blinded visual interpretation of a clinical diagnosis of the number of Normal-Scan and Abnormal-Scan Subjects who Converted to clinically probable Alzheimer's Disease (pAD).
Arm/Group | Not Clinically Probable Alzheimer's Disease | Clinically Probable Alzheimer's Disease
Number analyzed (Participants) | 143 | 81
Number of subjects
  Reader 1 - Normal | 111 | 31
  Reader 1 - Abnormal | 32 | 50
  Reader 2 - Normal | 72 | 21
  Reader 2 - Abnormal | 71 | 60
  Reader 3 - Normal | 108 | 37
  Reader 3 - Abnormal | 35 | 44
  Reader 4 - Normal | 98 | 28
  Reader 4 - Abnormal | 45 | 53
  Reader 5 - Normal | 98 | 29
  Reader 5 - Abnormal | 45 | 52
  Majority Reads - Normal | 98 | 29
  Majority Reads - Abnormal | 45 | 52

ADVERSE EVENTS:
Groups:
- Flutemetamol (18F) Injection: Flutemetamol (18F) Injection: All subjects will receive an intravenous dose of (18F) flutemetamol (less than 10 mg flutemetamol). The nominal activity of a single administration of (18F) flutemetamol will be 185 MBq.
Arm/Group | Flutemetamol (18F) Injection
Serious Adverse Events (participants affected / at risk) | 1/232
Other Adverse Events (participants affected / at risk) | 0/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flutemetamol (18F) Injection (N=232)
Anaphylactoid Reaction (Immune system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No